CLINICAL TRIAL: NCT01882556
Title: Is it Clinically Effective to Treat Arm Flexor Spasticity, With Botulinum Toxin - Type A (BoNTA) and Physiotherapy, as Soon as Signs of Abnormal Muscle Activity Are Observed?
Brief Title: Early Use of Botulinum Toxin in Spasticity Post Stroke.
Acronym: EUBoSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Collaborators: Keele University (Other); Stroke Research Network (Unknown)
Responsible Party: Principal Investigator, Cameron Lindsay, Mr, Sandwell & West Birmingham Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB-PG-0808-16319; 2010-021257-39 (EudraCT Number); ISRCTN57435427 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Stroke; Muscle Spasticity; Contracture
Keywords: Early treatment of spasticity.; Post stroke spasticity.
MeSH Terms: conditions — Stroke; Muscle Spasticity; Contracture | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin - Type A (onabotulinumtoxinA) (Experimental): Botulinum Toxin - Type A. One set of injections of up to 200 Units of Botox (Allergan). Injected to Biceps, Brachialis, Flexor Dig Superficialis, Flexor Dig Profundus, Flexor Carpi Radialis and Flexor Carpi Ulnaris.
  Interventions: Drug: onabotulinumtoxinA
- 0.9% NaCl Saline Injection (Placebo Comparator): Saline - Injected to Biceps, Brachialis, Flexor Dig Superficialis, Flexor Dig Profundus, Flexor Carpi Radialis and Flexor Carpi Ulnaris.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: onabotulinumtoxinA
  Other Names: Botox; Botulinum toxin type-A
  Arms: Botulinum Toxin - Type A (onabotulinumtoxinA)
Drug: Placebo
  Arms: 0.9% NaCl Saline Injection

SUMMARY:
Patients who survive a stroke are often left with an arm that cannot be used. One reason for this is that the muscles affected by the stroke become overactive. This is known as spasticity. Such unwanted muscle overactivity, if left untreated or poorly managed, can lead to limb deformities. For example, the wrist and fingers in the arm affected by spasticity become stiff and curl into a fist and the hand cannot be used for any functional purpose. Palm hygiene can become difficult and patients find this deformity unsightly and painful. Botulinum toxin (BT) has been shown to reduce muscle overactivity and is licensed for this purpose. In current practice this treatment is often used as a last line of defence. Although BT can reduce the muscle overactivity, when injected using current protocols, it seems to have little impact on the recovery of function and/or treating the limb deformities and pain. If BT can be given in the early stages of a stroke, i.e. as soon as the muscle overactivity is observed, then we will be able to treat spasticity and may prevent the limb deformities and pain from developing. We may also be able to assist the recovery of arm movement in some of the patients who would otherwise not have regained this. In addition to benefiting the patient, the prevention of secondary complications by early treatment may reduce the costs of long term care to the NHS . We hope to discover if our plan of providing early treatment with BT is more effective than the current approach. If we demonstrate that the treatment is effective we will be able to introduce this new method almost immediately within the NHS through our collaboration with doctors and therapists who are actively treating patients with this condition.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age.
2. Patients with stroke due to a primary cerebral haemorrhage/infarction, subarachnoid haemorrhage producing an upper motor syndrome affecting one body side which results in a hemiplegia
3. Capable of providing informed consent directly or indirectly, or, consent obtainable from next of kin or legal representative
4. No useful arm function (i.e. less than or equal to 2 on the grasp subsection of the Action Research Arm Test) at onset of spasticity

Exclusion Criteria:

1. Significant musculoskeletal conditions that affected upper limb function prior to the stroke
2. Unconscious or moribund during the screening period
3. Recovery of useful arm function (a score of 3 or more in the grasp section of the Action Research Arm Test) prior to injections
4. Patients with contraindications to electrical stimulation including active implants (e.g. cardiac assist devices), metal implants at site of stimulation, scar tissue/cancerous tissue at site of stimulation, uncontrolled epilepsy, deep vein thrombosis in limb / muscle being stimulated and pregnancy (or planned pregnancy)
5. Previous upper motor neurone syndrome or hypertonicity due to multiple sclerosis, spinal cord injury or other neurological disorder
6. Patients with a known hypersensitivity to any botulinum toxin or to any of the excipients of BOTOX® (i.e. Human serum albumin)
7. Patients with myasthenia gravis or Eaton Lambert Syndrome or other neuromuscular junction or myopathic disorder
8. Patients with infection at the proposed injection site(s)
9. Patients who are pregnant or may become pregnant at the time of the proposed injections and for the duration of the study
10. Current treatment with any antispasticity agent or previous injection with BOTOX

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test | 6 Months

SECONDARY OUTCOMES:
Spasticity | 6 Months
  In reducing focal spasticity in the arm as measured by surface electromyography (EMG) response of the wrist and elbow flexors to an externally imposed perturbation
Strength and Fatigue | 6 Months
  Strength and fatigue as measured by maximum isometric strength and the rate of force production in the wrist and elbow joints
Stiffness and passive range of movement. | 6 months
  Range of movement and force required to produce the same with a custom built device

OTHER OUTCOMES:
Quality of Life | 6 Months
  EuroQol EQ-5D
Care Giver Strain Index | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Anand D Pandyan, PhD, Study Chair — Keele University; Stephen G Sturman, MB ChB, Principal Investigator — SWBH NHS Trust
Locations (1):
- Sandwell and West Birmingham NHS Trust, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Background] Lindsay C, Simpson J, Ispoglou S, Sturman SG, Pandyan AD. The early use of botulinum toxin in post-stroke spasticity: study protocol for a randomised controlled trial. Trials. 2014 Jan 8;15:12. doi: 10.1186/1745-6215-15-12. PMID 24401159
- [Derived] Lindsay C, Humphreys I, Phillips C, Pandyan A. Estimating the cost consequence of the early use of botulinum toxin in post-stroke spasticity: Secondary analysis of a randomised controlled trial. Clin Rehabil. 2023 Mar;37(3):373-380. doi: 10.1177/02692155221133522. Epub 2022 Nov 3. PMID 36325678
- [Derived] Lindsay C, Ispoglou S, Helliwell B, Hicklin D, Sturman S, Pandyan A. Can the early use of botulinum toxin in post stroke spasticity reduce contracture development? A randomised controlled trial. Clin Rehabil. 2021 Mar;35(3):399-409. doi: 10.1177/0269215520963855. Epub 2020 Oct 11. PMID 33040610